CLINICAL TRIAL: NCT06418022
Title: Evaluating Fluid Responsiveness in Intensive Care Unit Patients Using VTI and Trendelenburg Positioning. TREND-US Trial.
Brief Title: Evaluating Fluid Responsiveness in ICU Patients Using VTI and Trendelenburg Positioning
Acronym: TREND-US
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lenox Hill Hospital (Other)
Responsible Party: Principal Investigator, Matthew Kheir, Principal Investigator, Lenox Hill Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-0441
Record Dates: First submitted 2024-05-06; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Shock; Fluid Overload; Cardiac Output, Low
Keywords: fluid; responsiveness; VTI; ICU; POCUS; ultrasound; Trendelenburg
MeSH Terms: conditions — Shock; Edema; Cardiac Output, Low

STUDY DESIGN:
Intervention Model Description: This is a single-center, minimal risk study that will include a total of 400 critically ill patients, aged 18 and older, that require fluid administration.
  In prior studies, fluid responsiveness has been shown after an IV fluid bolus with ≥15% increase in VTI or after a passive leg raise (PLR) with ≥ 15% increase in VTI. Similar to the other maneuvers such as the PLR maneuver, we hope to find an optimal cutoff in the increase in VTI after Trendelenburg positioning based on ROC analysis, with an increase of VTI >15% in patients after receiving IV fluids as the gold standard. There will be no intervention arm and patients will serve as their own control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Fluid challenge (control) (Other): This study is evaluating the potential of Trendelenburg positioning (TP) in determining fluid responsiveness by using the change in velocity time integral (VTI), and echocardiographic parameter that can be used as a surrogate for stroke volume and cardiac output.
  There are essentially two arms, whereby the patients is being compared to themselves.
  The "control arm" is the patient receiving a fluid challenge (FC; IV fluid bolus of 500cc crystalloids- either 0.9% Normal Saline or Lactated Ringer's solution) that the clinician would have given regardless of the study; the change of VTI is collected after administration of IV fluids with comparison to the baseline supine position.
  The "intervention arm" is the same patient undergoing TP from the baseline supine position to determine the change in VTI after subjecting to TP.
  Interventions: Device: Trendelenburg positioning VTI

INTERVENTIONS:
Device: Trendelenburg positioning VTI — There are essentially two arms, whereby the patients is being compared to themselves. The "intervention arm" is the same patient undergoing TP from the baseline supine position to determine the change in VTI after subjecting to TP.
  We will be using a Sonosite PX ultrasound system, which is intended for diagnostic ultrasound imaging or fluid flow analysis of the human body and, more specifically, for our echocardiographic measurements of velocity time integral (VTI; surrogate for stroke volume and cardiac output). The Sonosite PX is a general-purpose ultrasound system intended for use by qualified physicians and healthcare professionals, for evaluation by ultrasound imaging or fluid flow analysis of the human body. This is an FDA-cleared (510K# K200964) commercial device legally marketed in the United States that is being used in accordance with labeling.

SUMMARY:
Fluid administration is a commonly performed in the ICU for critically ill patients. However, it can lead to complications such as fluid overload, pulmonary edema, and increased mortality in some patients. Therefore, identifying patients who are likely to respond to fluid therapy is crucial for optimizing their management. Several methods have been used to assess fluid responsiveness, such as passive leg raising, stroke volume variation, and cardiac output monitoring. However, these methods have limitations and may not be feasible in all patients. In this study, the investigators aim to evaluate the use of velocity time integral (VTI) and Trendelenburg positioning in predicting fluid responsiveness in ICU patients.

DETAILED DESCRIPTION:
The investigators will perform an echocardiogram both in the supine and Trendelenburg positions for research purposes prior to the ICU team assessing fluid responsiveness (see paragraph below).

Critically ill patients in which fluid responsiveness is unclear typically admitted to the ICU routinely undergo a bedside echocardiogram in the supine position and then another echocardiogram still in the supine position after receiving IV fluids to assess the patient's fluid responsiveness (i.e., whether giving a small IV fluid bolus increases cardiac output). VTI is an echocardiographic surrogate for cardiac output and is routinely used in the ICU setting in addition to providing additional information on whether a patient is fluid responsive. This method is already standard practice in the medical and surgical ICU in our PCCM department.

Unfortunately, administering IV fluids can potentially cause adverse events such as pulmonary edema, heart failure, interstitial edema, respiratory failure, and death. The use of a method, such as the passive leg raise maneuver (i.e., raising patient's legs by 30 degrees for 1 minute and then evaluating hemodynamic measurements), help predict whether a patient would benefit from IV fluids prior to giving them fluids in order to prevent these aforementioned adverse events since it is a reversible process. Literature and current practice support the use of the passive leg raise (PLR) maneuver in predicting fluid responsiveness, where an increase of at least 15% signifies a positive fluid response. Similar to IV fluids, the PLR maneuver can cause adverse events, is cumbersome, and not feasible in certain circumstances. There is recent research which suggests that Trendelenburg positioning (TP) can be used as an alternative approach that is potentially safer and less cumbersome. This study aims to evaluate a cutoff increase in VTI that would be accurate in predicting fluid responsiveness in patients undergoing TP. As stated above, in our study we will see if placing the patient in TP (i.e., tilt head of the bed 15 degrees downward) will predict if the patient is fluid responsive. The investigators want use ROC analysis to determine the cutoff VTI increase and the accuracy of using TP in predicting fluid responsiveness. The gold standard is to check VTI prior to and after administering an IV fluid bolus and the current literature demonstrates that a VTI increase by 15% is indicative of an appropriate fluid response.

The patients in the study in the ICU will receive IV fluids regardless of our study based on the clinician's discretion (i.e., our study will not affect the decision of the clinician in any way). The bedside echocardiogram takes less than 2 minutes to perform and will not delay care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) admitted to the medical or surgical ICU.
* Patients who require fluid administration for suspicion of hypovolemia or indicated for volume expansion due to any one of the following: hypotension (systolic blood pressure < 90 mm Hg or mean arterial pressure < 65 mm Hg), tachycardia (heart rate > 100 beats per min), blood lactate > 2.0 mmol/L, skin mottling, oliguria (urine output < 30 ml/hr), or requiring vasopressor/inotrope support.
* Patients who are able to tolerate the Trendelenburg position.

Exclusion Criteria:

* Pregnancy.
* Prisoners and institutionalized patients.
* Patients who are not able to tolerate the Trendelenburg position. This includes patients with increased intra-cranial hypertension, intra-abdominal hypertension and gastric retention which places a risk for stomach fluid aspiration.
* Unsatisfactory cardiac echogenicity (an inability to correctly align the Doppler beam to generate reliable VTI measurements at the left ventricular outflow tract [LVOT]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in VTI cutoff in TP that predicts fluid responsiveness | ~1 year
  The objective of this study is to determine the change in VTI cutoff with Trendelenburg positioning that would predict fluid responsiveness in medical and surgical intensive care unit patients.

SECONDARY OUTCOMES:
Determine if patient factors are independently associated with fluid responsiveness | ~1 year
  Evaluate other patient factors (e.g., demographics) to determine if they are independently associated with fluid responsiveness.
Association of Trendelenburg positioning on the effect on hemodynamic parameters | ~1 year
  Evaluate the effect of Trendelenburg positioning (TP) and fluid challenge (FC) on hemodynamic parameter of blood pressure (i.e., if there is a statistically significant change in the hemodynamic parameter after TP or FC).
Association of Trendelenburg positioning on the effect on hemodynamic parameters | ~1 year
  Evaluate the effect of Trendelenburg positioning (TP) and fluid challenge (FC) on hemodynamic parameter of heart rate (i.e., if there is a statistically significant change in the hemodynamic parameter after TP or FC).
Association of Trendelenburg positioning on the effect on hemodynamic parameters | ~1 year
  Evaluate the effect of Trendelenburg positioning (TP) and fluid challenge (FC) on hemodynamic parameter of pulse pressure (i.e., if there is a statistically significant change in the hemodynamic parameter after TP or FC).
Association of Trendelenburg positioning on the effect on hemodynamic parameters | ~1 year
  Evaluate the effect of Trendelenburg positioning (TP) and fluid challenge (FC) on hemodynamic parameter of central venous pressure (i.e., if there is a statistically significant change in the hemodynamic parameter after TP or FC).
Evaluate the predictive accuracy of the change in VTI versus other hemodynamic parameters | ~1 year
  Use receiver operating characteristic (ROC) curves to compare the predictive accuracy of the change in VTI compared to the change of certain hemodynamic parameters (e.g., pulse pressure, systolic blood pressure, diastolic blood pressure) with Trendelenburg positioning.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kheir, MD, Principal Investigator — Lenox Hill Hospital- Northwell Health
Locations (1):
- Lenox Hill Hospital- Northwell Health, New York, New York, United States